CLINICAL TRIAL: NCT03010748
Title: Multi-center Clinical Trial on Corneal Morphology Analysis in Chinese Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Eye Hospital (Other)
Collaborators: Jilin University (Other); Xi'an Jiaotong University (Other); Second People's Hospital of Yunnan Province (Other); Wuhan General Hospital of Guangzhou Military Command (Other); Xinjiang Medical University (Other); Gansu Provincial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Tianjin EH-pentacam
Record Dates: First submitted 2016-12-28; First posted 2017-01-05 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Cornea
Keywords: corneal morphology; Chinese population; corneal curvature; corneal thickness; higher order aberrations
MeSH Terms: conditions — Corneal Diseases | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chinese population: Chinese population of different nation from several provinces.
  Interventions: Device: Scheimpflug tomography system (Pentacam) measurement

INTERVENTIONS:
Device: Scheimpflug tomography system (Pentacam) measurement — The Scheimpflug tomography system (Pentacam,Oculus GmbH, Wetzlar, Germany) is a rotating Scheimpflug camera that measures 138,000 true elevation points to compute corneal topography. Patients were asked to blink twice and then look at the fixation device. Image acquisition was a 2-second scan of 50 rotational Scheimpflug images through the corneal sighting point, the point where the ray of light from the fovea to the fixation device crossed the cornea. All measurements were performed just after a blink to minimize the effect of tear film alteration on the data. Acceptable maps had at least 10.0 mm of corneal coverage with no extrapolated data in the central 9.0 mm zone.

SUMMARY:
Based on the corneal morphometry instrumentation Oculus Pentacam, which is commonly used before and after clinical refractive surgery, we will collect the corneal morphological and biologic parameters of the population under refractive surgery screening in refractive surgery centers around the country, and construct corneal morphology database in different living areas of Chinese people. Based on this, compared with the suspected keratoconus and keratoconus population, the screening criteria and reference standards accord with the characteristics of keratoconus of Chinese ethnic will be achieved.

DETAILED DESCRIPTION:
The safety of refractive surgery has always been the focus of attention, keratoconus screening is the most important part for the preoperative examination of refractive surgery. Favorable tools and appropriate indicators are the premise of fast and accurate screening, and the corneal morphology from various regions of China have various characteristics, the use of uniform standards developed by foreign screening will always induce a lot of problems, for example, the differences of cornea morphological features between European and American ethnic and Chinese race, as well as the corneal morphometric indicators between various regions of China, will cause varying degrees of false-positive or false-negative screening results. Based on this, in order to further improve the safety of refractive surgery effectively and to obtain the effective and accurate screening of suspected keratoconus population, this study will be conducted to collect the corneal morphological characteristics database of Chinese people from all over the country, and to develop a database of Chinese ethnographic characteristics for screening keratoconus indicators and reference valuable to guide clinical screening and surgical design.

ELIGIBILITY:
Inclusion Criteria:

* No less than 18 years old, in good health, have no active disease in the body and eye, have permanent resident status and have lived in the local area for at least 5 years (please mark the nation).

Exclusion Criteria:

* Eye diseases, glaucoma, ocular hypertension, glaucoma patients with normal pressure, fundus lesions, ptosis and other eyelid abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese population of different nation from several provinces,including Jilin, Xi'an, Yunnan, Wuhan,etc.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2015-11; Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
corneal thickness | preoperative

SECONDARY OUTCOMES:
corneal curvature measured by the Pentacam system | preoperative
coma aberration measured by the Pentacam system | preoperative
aspherical index measured by the Pentacam system | preoperative
spherical aberration measured by the Pentacam system | preoperative
corrected distance visual acuity | preoperative
uncorrected distance visual acuity | preoperative
refractive diopter | preoperative
corneal volume measured by the Pentacam system | preoperative
kapple angle measured by the Pentacam system | preoperative
introcular pressure | preoperative
corneal diameter measured by the Pentacam system | preoperative
anterior chamber depth measured by the Pentacam system | preoperative
anterior chamber angle measured by the Pentacam system | preoperative

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, director, Study Director — Tianjin Eye Hospital; Xiaoyu li, Principal Investigator — Second People's Hospital of Yunnan Province; Yan Zhang, Principal Investigator — Jilin University; Jun Yang, Principal Investigator — Gansu Provincial Hospital; Jing Li, Principal Investigator — Xi'an Jiaotong University; Xianglong Yi, Principal Investigator — Xinjiang Medical University; Zhengwei Shen, Principal Investigator — Wuhan General Hospital of Guangzhou Military Command
Locations (1):
- Tianjin Eye Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silverman RH, Urs R, RoyChoudhury A, Archer TJ, Gobbe M, Reinstein DZ. Combined tomography and epithelial thickness mapping for diagnosis of keratoconus. Eur J Ophthalmol. 2017 Mar 10;27(2):129-134. doi: 10.5301/ejo.5000850. Epub 2016 Aug 8. PMID 27515569
- [Background] Chan TCY, Biswas S, Yu M, Jhanji V. Comparison of corneal measurements in keratoconus using swept-source optical coherence tomography and combined Placido-Scheimpflug imaging. Acta Ophthalmol. 2017 Sep;95(6):e486-e494. doi: 10.1111/aos.13298. Epub 2016 Nov 2. PMID 27805316
- [Background] Patrao LF, Canedo AL, Azevedo JL, Correa R, Ambrosio R Jr. Differentiation of mild keratoconus from corneal warpage according to topographic inferior steepening based on corneal tomography data. Arq Bras Oftalmol. 2016 Jul-Aug;79(4):264-7. doi: 10.5935/0004-2749.20160075. PMID 27626155
- [Background] Naderan M, Rajabi MT, Zarrinbakhsh P, Farjadnia M. Is keratoconus more severe in pediatric population? Int Ophthalmol. 2017 Oct;37(5):1169-1173. doi: 10.1007/s10792-016-0382-5. Epub 2016 Oct 25. PMID 27783185
- [Derived] Ma J, Zhao L, Yang Y, Yun D, Yu-Wai-Man P, Zhu Y, Chen C, Li JO, Li M, Zhang Y, Cui T, Meng X, Zhang L, Zhang J, Song Y, Lei Y, Liu J, Huangfu X, Jiang L, Cai J, Wu H, Shang L, Wen D, Yi X, Zhang Y, Li X, Xiao J, He R, Yang Y, Yang J, Cheng GPM, Bai J, Zhong X, Guo H, Yan P, Wang Y, Lin H. Associations Between Regional Environment and Cornea-Related Morphology of the Eye in Young Adults: A Large-Scale Multicenter Cross-Sectional Study. Invest Ophthalmol Vis Sci. 2021 Feb 1;62(2):35. doi: 10.1167/iovs.62.2.35. PMID 33620373
- See also: Combined tomography and epithelial thickness mapping for diagnosis of keratoconus. — http://www.eur-j-ophthalmol.com/article/640efc2c-7e6d-47ad-b8ca-19ef814a8101
- See also: Comparison of corneal measurements in keratoconus using swept-source optical coherence tomography and combined Placido-Scheimpflug imaging — http://onlinelibrary.wiley.com/doi/10.1111/aos.13298/abstract;jsessionid=B34D7E065EA943A24C0B230AE3875DDD.f02t03
- See also: Differentiation of mild keratoconus from corneal warpage according to topographic inferior steepening based on corneal tomography data — http://www.scielo.br/scielo.php?script=sci_arttext&pid=S0004-27492016000400264&lng=en&nrm=iso&tlng=en
- See also: Is keratoconus more severe in pediatric population? — http://link.springer.com/article/10.1007%2Fs10792-016-0382-5